CLINICAL TRIAL: NCT00675506
Title: Physiologic Effects of Long-Term GHRH1-44 in Abdominal Obesity
Brief Title: Effectiveness of Growth Hormone Releasing Hormone in Reducing Abdominal Fat in People Who Are Obese
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 574; 1R01HL085268-01A1 (NIH)
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Results first posted 2013-01-07 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Abdominal Obesity; Growth Hormone Deficiency
Keywords: Growth Hormone Releasing Hormone; Growth Hormone Pulse; Visceral Adipose Tissue; Carotid Intima-Media Thickness
MeSH Terms: conditions — Obesity, Abdominal; Dwarfism, Pituitary | interventions — Growth Hormone-Releasing Hormone; tesamorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive treatment with growth hormone releasing hormone 1-44 (TH9507).
  Interventions: Drug: Growth hormone releasing hormone (GHRH) 1-44
- 2 (Placebo Comparator): Participants will receive treatment with placebo medication.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Growth hormone releasing hormone (GHRH) 1-44 — 2-mg sub-cutaneous injections once daily for 12 months
  Other Names: TH9507
  Arms: 1
Drug: Placebo — 2-mg sub-cutaneous injections once daily for 12 months
  Arms: 2

SUMMARY:
Obesity, a condition that occurs when a person has too much body fat, affects about 31% of people in the United States. It is associated with increased risk of diabetes, high blood pressure, high cholesterol, and cardiovascular disease. Abdominal obesity, in particular, is also associated with low levels of growth hormone, a hormone that affects rate of growth and the way the body uses energy. Growth hormone releasing hormone (GHRH) is a substance that makes the body naturally increase its own growth hormone levels. Administering GHRH to people who are obese may help return their growth hormone levels to normal and, in turn, may lead to reduced abdominal fat and improved cardiovascular function. This study will evaluate the effectiveness of synthetic GHRH in decreasing the amount of abdominal fat and improving cardiovascular function in people who are obese.

DETAILED DESCRIPTION:
Obesity, defined as having a high amount of excess body fat, is one of the most wide-spread health problems of today. A variety of factors can lead to obesity. These factors include physical inactivity, family history and genetics, metabolism, and hormone imbalance. The excess body fat in obesity increases a person's risk of a number of life-threatening diseases, including heart disease, gall stones, type 2 diabetes, and certain types of cancer. People with abdominal obesity, where fat is stored predominantly around a person's midsection, are particularly prone to weight-related diseases. Studies have shown that administration of growth hormone to obese people reduces abdominal fat, but can be associated with adverse side effects. GHRH is a natural hypothalamic peptide that stimulates growth hormone release. GHRH may be able to normalize growth hormone levels, reduce abdominal fat, and lessen risk for cardiovascular disease in people who are obese, without the associated side effects of growth hormone administration. However, further study is needed on GHRH. This study will evaluate the safety and effectiveness of synthetic GHRH in decreasing the amount of abdominal fat and improving cardiovascular function in people who are obese.

Participation is this study will last 1 year from screening and will include 9 study visits. During Visit 1, participants will undergo screening tests that will include a medical history, a physical exam, body measurements, a blood draw, a urine test, a GHRH+Arginine stimulation test, an electrocardiogram (ECG), and a test for the presence of blood in stool. Eligible participants will return within the next 3 weeks for an inpatient clinic stay for Visit 2. Participants will be asked to keep a food record of all food consumed during the 4 days before the second visit. Visit 2 will include a physical exam, a medical and smoking history, a review of current medications, body measurements, an overnight blood draw, a body metabolism evaluation, an oral glucose tolerance test, and two questionnaires. Also during Visit 2, participants will be assigned randomly to treatment with active GHRH or placebo. Participants will then be taught how to give themselves injections of the study drug, which will be taken daily for 12 months. Participants will also receive a 1-month supply of study drug and will be supplied with refills in subsequent study visits. Upon starting treatment, participants will undergo more testing, including a whole body DEXA scan, abdominal computed tomography (CT) scan, carotid ultrasound, and ECG.

Visit 3 will occur at Week 2 of treatment and will include a review of study medications, questions about any side effects experienced, vital sign measurements, a blood draw, an ECG, and, if female, a urine test. Visits 4, 5, and 7 will be identical to Visit 3 and will occur at Months 1, 3, and 9 respectively. Visit 6 will occur at Month 6 and will be identical to Visit 2 but without the overnight blood draw. Visit 8 will occur at Month 12 and will be identical to Visit 2, except no further study drug will be dispensed. At Month 13, participants will complete the final study visit, which will include repeat tests from Visit 1.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) greater than or equal to 30 kg/m2
* Waist circumference greater than or equal to 102 cm in men and greater than or equal to 88 cm in women
* Relative growth hormone (GH) deficiency, defined as a peak GH value of less than or equal to 8 ng/mL on Arginine-GHRH stimulation test
* Hemoglobin level greater than 12.0 g/dL
* Serum glutamic oxaloacetic transaminase and serum glutamic pyruvic transaminase less than 2.5 times the upper limit of normal
* Creatinine level less than 1.5 mg/dL
* Follicle stimulating hormone less than 20 IU/L in women
* Negative mammogram within 1 year of study entry for women older than 40 years of age

Exclusion Criteria:

* Obesity due to a known secondary cause (e.g., Cushing's syndrome, hypothyroidism) or a history of gastric bypass procedure
* Known hypersensitivity to GHRH 1-44 (TH9507)
* Known history of diabetes, fasting blood sugar less than 125 mg/dL, or antidiabetic drug use
* Using any weight lowering drugs
* Using estrogen, hormone replacement therapy, oral contraceptives, testosterone, glucocorticoids, anabolic steroids, GHRH, GH, or insulin-like growth factor-1 (IGF-1) within 3 months of study entry
* Changes in lipid lowering or antihypertensive regimen within 3 months of study entry
* Long-term illness, including anemia, chronic kidney disease, and liver disease
* History of cancer (except patients with surgically cured basal cell or squamous cell skin cancers) or history of abnormalities on age appropriate malignancy screen, including mammography, colonoscopy, and prostate exam (or prostate specific antigen greater than 5 ng/mL)
* History of hypopituitarism, pituitary surgery, pituitary/brain radiation, traumatic brain injury, or any other condition known to affect the growth hormone axis
* History of any recent cardiovascular event, including heart attack, stroke, transient ischemic attack, unstable angina pectoris, or oxygen-dependent severe pulmonary disease, within 3 months of study entry
* Clinical depression or other psychiatric illness that will not allow completion of the study as per investigator's judgement
* History of or current eating disorder
* History of recent alcohol or substance abuse (less than 1 year before study entry)
* Positive pregnancy test or breastfeeding females and positive fecal occult blood test
* Women of childbearing potential not currently using nonhormonal birth control methods, including barrier methods (e.g., IUD, condoms, diaphragms) or abstinence
* Currently enrolled in another investigational device or drug trial(s) or has received other investigational agent(s) within 28 days of study entry
* Any condition that would make this clinical trial detrimental to the patient, as judged by the patient's physician
* History of noncompliance with other therapies
* Any condition in which compliance with the study protocol is unlikely

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven K. Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Stanley TL, Feldpausch MN, Murphy CA, Grinspoon SK, Makimura H. Discordance of IGF-1 and GH stimulation testing for altered GH secretion in obesity. Growth Horm IGF Res. 2014 Feb;24(1):10-5. doi: 10.1016/j.ghir.2013.11.001. Epub 2013 Nov 15. PMID 24291224
- [Derived] Makimura H, Murphy CA, Feldpausch MN, Grinspoon SK. The effects of tesamorelin on phosphocreatine recovery in obese subjects with reduced GH. J Clin Endocrinol Metab. 2014 Jan;99(1):338-43. doi: 10.1210/jc.2013-3436. Epub 2013 Dec 20. PMID 24178787
- [Derived] Makimura H, Feldpausch MN, Rope AM, Hemphill LC, Torriani M, Lee H, Grinspoon SK. Metabolic effects of a growth hormone-releasing factor in obese subjects with reduced growth hormone secretion: a randomized controlled trial. J Clin Endocrinol Metab. 2012 Dec;97(12):4769-79. doi: 10.1210/jc.2012-2794. Epub 2012 Sep 26. PMID 23015655

RESULTS

PARTICIPANT FLOW:
Groups:
- TH9507: Participants received treatment with growth hormone releasing hormone 1-44 (TH9507).
  Growth hormone releasing hormone (GHRH) 1-44 : 2-mg sub-cutaneous abdominal injections once daily for 12 months
- Placebo: Participants received treatment with placebo medication.
  Placebo : 2-mg sub-cutaneous abdominal injections once daily for 12 months
Period: Overall Study
Arm/Group | TH9507 | Placebo
Started | 31 | 29
Received Intervention | 29 (Two subjects did not start treatment: 1) disclosed cancer history, 2) declined participation.) | 29
Completed | 19 | 17
Not Completed | 12 | 12
Not completed — Lost to Follow-up | 1 | 5
Not completed — Lost interest | 3 | 5
Not completed — Elevated fasting glucose | 2 | 1
Not completed — Elevated IGF-1 prior to treatment | 1 | 0
Not completed — Elevated IGF-1 | 2 | 0
Not completed — Hypersensitivity Reaction | 1 | 0
Not completed — Disclosed history of cancer | 1 | 0
Not completed — Declined participation | 1 | 0
Not completed — Schedule conflict | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received treatment with placebo medication.
  Placebo: 2-mg sub-cutaneous abdominal injections once daily for 12 months
- Total: Total of all reporting groups
Arm/Group | TH9507 | Placebo | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 29 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (7.1) | 39.9 (9.5) | 41.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 20 | 19 | 39
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Visceral Adipose Tissue Volume
Description: Abdominal visceral adipose tissue and subcutaneous adipose tissue were assessed using a single crosssectional slice from noncontrast computed tomography at the L4 level. The change in abdominal visceral adiposity between baseline and twelve months is reported.
Time Frame: Measured at baseline and Months 6 and 12
Population: All data were included in the analysis by intention to treat principle. For participants who did not complete a 12-month visit, last observation carried forward was performed for those participants for whom interim data post the baseline visit was available. Data from 6 month is utilized in the linear mixed effects modeling.
Measure: Mean (Standard Error); unit: cm2
Groups:
- TH9507: Participants received treatment with growth hormone releasing hormone 1-44 (TH9507).
  TH9507: Growth hormone releasing hormone (GHRH) 1-44 : 2-mg sub-cutaneous abdominal injections once daily for 12 months.
Arm/Group | TH9507 | Placebo
Number analyzed (Participants) | 29 | 29
cm2 | -16 (9) | 19 (9)

2. Secondary Outcome: Change in Carotid Intima-media Thickness
Description: Carotid intima media thickness imaging of the common carotid artery was conducted using a high-resolution 7.5-MHz phased-array transducer (SONOS 2000/2500. The change of the carotid intima media thickness measurement between baseline and 12 months is reported.
Time Frame: Measured at baseline and Months 6 and 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mm
Arm/Group | TH9507 | Placebo
Number analyzed (Participants) | 29 | 29
mm | -0.03 (0.01) | 0.01 (0.01)

3. Secondary Outcome: Change in Lipid Profile (Total Cholesterol, High-density Lipoproteins [HDL] Cholesterol, Low-density Lipoproteins [LDL] Cholesterol, Triglycerides)
Description: Lipid Profile (total cholesterol, high-density lipoproteins [HDL] cholesterol, low-density lipoproteins [LDL] cholesterol, triglycerides)was determined after an overnight fast. The change in lipid profile between baseline and 12 months is reported.
Time Frame: Measured at baseline and Months 6 and 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | TH9507 | Placebo
Number analyzed (Participants) | 29 | 29
mg/dL
  Total Cholesterol | 4 (4) | 7 (5)
  High-density lipoproteins [HDL] cholesterol | 4 (1) | 3 (1)
  Low-density lipoproteins [LDL] cholesterol | 4 (4) | 1 (4)
  Triglycerides | -26 (16) | 12 (8)

4. Secondary Outcome: Change in Glucose Tolerance as Measured by Oral Glucose Tolerance Test
Description: Glucose tolerance was determined after an overnight fast using standard 75 gram oral glucose tolerance test (OGTT) with glucose measured at timepoints 0, 30, 60, 90 and 120. Change in glucose tolerance (fasting and 2 hour OGTT) between baseline and twelve months is reported.
Time Frame: Measured at baseline and Months 6 and 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | TH9507 | Placebo
Number analyzed (Participants) | 29 | 29
mg/dL
  Fasting Glucose | 2 (3) | 1 (2)
  2 Hour OGTT Glucose | -11 (7) | -3 (8)

5. Secondary Outcome: Change in Growth Hormone Pulse Characteristics (Median Pulse Mass) as Assessed by Overnight Frequent Sampling of Growth Hormone
Description: Overnight frequent sampling of growth hormone levels was performed and characteristics of pulsatile secretion were determine using automated deconvolution (using AutoDecon software). Based on the deconvolution, the median pulse mass (in nanograms per millileter of growth hormone) was calculated. A positive number indicates an increase in median pulse mass between baseline and 12 months.
Time Frame: Measured at baseline and Month 12
Population: All available data (all participants for whom change from baseline to 12 months was available)
Measure: Mean (Standard Deviation); unit: nanograms/milliliter
Arm/Group | TH9507 | Placebo
Number analyzed (Participants) | 18 | 12
nanograms/milliliter | 0.54 (1.35) | 0.20 (0.30)

6. Secondary Outcome: Mitochondrial Function (Post-exercise Phosphocreatine Recovery [ViPCr]) by 31P-MRS
Description: Change in post-exercise phosphocreatine recovery [ViPCr] between baseline and 12 months (positive change indicates increase in the variable between baseline and 12 months). ViPCR is the initial rate of phosphocreatine recovery normalized based on participant effort. Greater ViPCr represents relatively better mitochondrial function.
Time Frame: Measured at Baseline and Month 12
Population: All available data. Assessment of mitochondrial function could not be performed in all patients.
Measure: Mean (Standard Deviation); unit: milliMoles/second
Arm/Group | TH9507 | Placebo
Number analyzed (Participants) | 9 | 11
milliMoles/second | 0.01 (11.3) | -1.02 (5.7)

ADVERSE EVENTS:
Time Frame: Safety visits occurred at 2 weeks, 1, 3, 6 and 9 months at which time fasting glucose and IGF-1 were monitored.
Arm/Group | TH9507 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 28/31 | 26/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TH9507 (N=31) | Placebo (N=29)
Injection site bruising (Skin and subcutaneous tissue disorders) | 17 (17) | 21 (21)
Hypertension (Cardiac disorders) | 8 (8) | 5 (5)
Injection-site bleeding (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)
Injection-site pain (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Tingling/ Paresthesia (Nervous system disorders) | 3 (3) | 1 (1)
Peripheral edema (Vascular disorders) | 3 (3) | 1 (1)
Injection site puritis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Injection site erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Atypical chest pain (Psychiatric disorders) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Fatigue (Nervous system disorders) | 2 (2) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 5 (5)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Mechanical injury (General disorders) | 0 (0) | 3 (3)
Musculoskeletal injury (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 6 (6)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Toothache (General disorders) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No